CLINICAL TRIAL: NCT06477653
Title: A Pilot Phase 2 Study of the Safety and Efficacy of Dupilumab as Add-on Therapy for Hypereosinophilic Syndrome With Partial Clinical Response to Eosinophil-Depleting Biologic Agents
Brief Title: Dupilumab as Add-On Therapy for Hypereosinophilic Syndrome With Partial Clinical Response to Eosinophil-Depleting Biologic Agents
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001979; 001979-I
Record Dates: First submitted 2024-06-26; First posted 2024-06-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12-03

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Hypereosinophilic Syndrome; Eosinophil; Monoclonal Antibody; Clinical Trial; Treatment
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dupilumab in addition to mepolizumab, reslizumab, or benralizumab (at least 24 but up to 48 weeks) (Experimental): Dosing for an individual will be determined based on the nature of their residual symptoms and the FDA-approved dosing for that indication. Patients will self-administer using pre-filled syringes with needle shield or pre-filled pens. Patients with asthma and/or atopic dermatitis will receive a loading dose of 600 mg subcutaneously (followed by 300 mg SC every 2 weeks. Patients with Chronic Rhinosinusitis with Nasal Polyposis will not receive a loading dose and will be treated with 300 mg subcutaneously every 2 weeks. Patients with Eosinophilic Esophagitis will not receive a loading dose of 600 mg subcutaneously and will be treated with 300 mg subcutaneously weekly. Patients who meet criteria for more than one indication will be treated with the higher dose.
  Interventions: Biological: dupilumab

INTERVENTIONS:
Biological: dupilumab — Dupilumab is an interleukin-4 receptor alpha antagonist. Dosing for an individual will be determined based on the nature of their residual symptoms and the FDA-approved dosing for that indication.

SUMMARY:
Background:

Hypereosinophilic syndrome (HES) is a blood disorder that causes high levels of white blood cells called eosinophils. HES can damage the lungs and airways, intestines, skin, and other organs. The current primary treatment for HES can cause serious side effects. Secondary treatments do not work in all people.

Objective:

To test an approved drug (dupilumab), combined with other drugs, in people with HES.

Eligibility:

People aged 18 years and older who take drugs (mepolizumab, reslizumab, or benralizumab) to treat HES.

Design:

Participants will have up to 6 clinic visits and 7 remote visits in up to 48 weeks.

Participants will be screened. They will have blood and urine tests. They will have a test of their heart function. They will take surveys about how HES affects their daily life. Some participants may have a bone marrow biopsy: A sample of tissue and fluid from inside a bone will be removed with a large needle.

Participants will have other tests specific to their symptoms. For example, those with symptoms affecting their lungs will have breathing tests. Others may have tests that target symptoms in their sinuses, gastrointestinal tract, or skin.

Dupilumab is injected under the skin once every 1 or 2 weeks. Dose and timing will vary among participants. They will be taught how to inject themselves at home between clinic visits. They will take dupilumab plus their current medications for 24 weeks. If the drug is helping them, they will continue taking it for another 24 weeks.

Participants will have a final visit 12 weeks after their last dose.

DETAILED DESCRIPTION:
Study Description:

The purpose of this study is to evaluate the efficacy and tolerability of dupilumab in reducing clinical manifestations in patients with hypereosinophilic syndrome (HES) and persistent eosinophil-related pulmonary, skin, gastrointestinal, or sinus symptoms despite eosinophil reduction in response to eosinophil-lowering biologic therapy. Patients who meet criteria for HES and are currently receiving mepolizumab, reslizumab or benralizumab with persistent symptoms (as above) despite absolute eosinophil count (AEC)<0.5x10^9/L will be eligible to enroll. Participants will be treated with dupilumab at the US Food and Drug Administration (FDA)-approved doses for asthma, atopic dermatitis, chronic rhinosinusitis with nasal polyposis (CRSwNP), or eosinophilic esophagitis (EoE) depending on their residual symptoms Participants will have clinical evaluations and AEC measured every 4 weeks for 24 weeks. Participants who remain in clinical remission and have an AEC<0.5x10^9/L will be eligible to continue dupilumab therapy for an additional 24 weeks with tapering of background therapy (other than the eosinophil-lowering biologic) as clinically tolerated.

Objectives:

Primary Objective: To assess the efficacy of add-on dupilumab therapy in reducing residual pulmonary, skin, esophageal, and sinus symptoms in patients with HES in complete hematologic and partial clinical remission on eosinophil-lowering biologics

Secondary Objective: To determine the effect of eosinophil-lowering therapy on dupilumab-induced blood eosinophilia and eosinophil-associated AEs

Endpoints:

Primary Endpoint: Clinical improvement on dupilumab therapy at 24 weeks, as assessed by HES-Most Bothersome Symptom (HES-MBS) and HES-Symptom Inventory (HES-SI)

Secondary Endpoints:

1. Incidence of new or worsening symptoms or signs attributable to eosinophilia requiring therapeutic intervention through week 24
2. Peripheral blood AEC at 4, 12, and 24 weeks.
3. Proportion of patients who maintain an eosinophil count below 0.5x10^9/L at 4, 12 and 24 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Age >=18 years
2. Documented diagnosis of HES with historic AEC>1.5x10^9/L on two occasions, no secondary etiology for the eosinophilia despite careful clinical evaluation, and evidence of end organ damage (histologic evidence of tissue infiltration by eosinophils and/or objective evidence of clinical pathology in any organ system that is temporally associated with eosinophilia and not clearly attributable to another cause)
3. Currently receiving treatment with an eosinophil-lowering biologic (mepolizumab, reslizumab, or benralizumab) for a minimum of 24 weeks
4. AEC<0.5x10^9/L
5. Residual symptoms after a minimum of 24 weeks of eosinophil-lowering biologic therapy with at least 1 most bothersome symptom of moderate severity (HES-SI score >=2) consistent with >=1 of the following diagnoses:

   a. asthma, defined as physician-documented asthma requiring medium to high dose inhaled corticosteroids + long-acting beta agonist b. atopic dermatitis, defined as physician-documented chronic or recurrent inflammatory skin disease

   c. CRSwNP, defined as evidence of rhinosinusitis and nasal polyposis on physical examination or imaging

   d. EoE, defined as biopsy-proven esophageal eosinophilia >15 eosinophils/high power field
6. For participants who can become pregnant: sexual abstinence or use of highly effective contraception (i.e., partner vasectomy, bilateral tubal ligation, IUD, progestin implants, and other hormonal methods) starting 4 weeks prior to study drug initiation and agreement to use such a method during study participation and for an additional 12 weeks after the end of study drug administration
7. Participation in NIH protocol 94-I-0079 (Activation and function of eosinophils in conditions with blood or tissue eosinophilia)
8. Ability of subject to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or lactation
2. Known allergic reaction to dupilumab or any of the excipients in Dupixent(TM)
3. Febrile illness within 7 days of enrollment
4. Treatment with an investigational drug or other intervention other than mepolizumab, reslizumab, or benralizumab within 12 weeks or 4 half-lives of the investigational agent (whichever is longer).
5. Known or suspected acquired or inborn immunodeficiency disorder, including HIV infection
6. Known diagnosis of eosinophilic granulomatosis with polyangiitis
7. Change in eosinophil-active therapy within the past 6 weeks, including but not limited to topical corticosteroids, leukotriene inhibitors, initiation or change of a food-elimination diet regimen or re-introduction of a previously eliminated food (in patients with gastrointestinal involvement), and proton pump inhibitors (in patients with gastrointestinal involvement)
8. Planned or anticipated major surgical procedure during the study
9. Active parasitic infection
10. History of malignancy within 5 years, excluding completely treated in situ carcinoma of the cervix, or squamous or basal cell carcinoma of the skin
11. Any condition that, in the investigator s opinion, places the patient at undue risk by participating in the study

For patients with eosinophilic gastrointestinal disease only:

1. Active infection with Helicobacter pylori
2. History of achalasia, Crohn s disease, ulcerative colitis, celiac disease, or prior esophageal surgery
3. Any esophageal stricture unable to be passed with a standard, diagnostic, 9 to 10 mm upper endoscope

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement on dupilumab therapy as assessed by HES-MBS (HES-most bothersome symptom) and HES-SI (HES-Symptom Inventory). | Baseline through week 24
  To assess the efficacy of add-on dupilumab therapy in reducing residual asthma, skin, esophageal, and sinus symptoms in patients with HES in complete hematologic and partial clinical remission on eosinophil-lowering biologics.

SECONDARY OUTCOMES:
Incidence of new or worsening symptoms or signs attributable to eosinophilia requiring therapeutic intervention. | During the first 24 weeks of study.
  To determine the effect of eosinophil-lowering therapy on dupilumab-induced blood eosinophilia and eosinophil-associated AEs.
Peripheral blood absolute eosinophil counts. | At 4, 12 and 24 weeks.
  To determine the effect of eosinophil-lowering therapy on dupilumab-induced blood eosinophilia and eosinophil-associated AEs.
Proportion of patients who maintain an eosinophil count below 0.5 x 10^9/L. | At 4, 12 and 24 weeks.
  To determine the effect of eosinophil-lowering therapy on dupilumab-induced blood eosinophilia and eosinophil-associated AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001979-I.html